CLINICAL TRIAL: NCT05630391
Title: Approach to the Coronavirus With Patient With High-Fidelity Simulation Training: A Mixed Method Study
Brief Title: High-Fidelity Simulation Training: A Mixed Method Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, özlem doğu, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Simcovid
Record Dates: First submitted 2022-10-17; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Simulation of Physical Illness; Satisfaction
Keywords: COVID-19; Simulation; Personal protective equipment; Nurse
MeSH Terms: conditions — Personal Satisfaction; COVID-19 | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the process of teaching personnel protective equipment (PPE) use with the scenario-based high-fidelity simulation mannikin, a simulation application was made with 26 students. The simulation scenario was implemented with 13 groups consisting of 3 students each playing different roles (nurse, head nurse, patient relative). Throughout the scenario, the students who played the role of the nurse and the head nurse simulated the PPE wearing-removal practice in a way to cover all steps of the process (preparation, implementation, and evaluation). During the implementation of the scenario, the student playing the role of the patient's relative provided guiding clues to the nurse when needed. Debriefing was started right after the simulation. Frequency of administration the implementation of each group is once and the debriefing stage where the learning process was reinforced and lasted 30 minutes.
  Interventions: Device: High-Fidelity Simulation Manikin
- Control (Other): The 26 students who constituted the control group performed the personnel protective equipment (PPE) wearing-removal practice once under the supervision of the researcher at the Fundamentals of Nursing skills laboratory. Frequency of administration the implementation of each group is once. The students applied experiential learning principles through active experience and reflective observation.
  Interventions: Other: Education

INTERVENTIONS:
Device: High-Fidelity Simulation Manikin — A high-fidelity simulator was developed to teach skills in nursing education, and it is sized to represent an adult male patient. The mannequin can be controlled using a computer program, it can breathe, and its vital signs can be monitored using a bedside monitor.
  Arms: Intervention
Other: Education — Training for 26 nursing students who constituted the control group performed personnel protective equipment (PPE) wearing-removal practice
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare in describe first-year nursing students' skills. The main questions it aims to answer are:

* Are nursing students who perform the simulation practice with the scenario-based high-fidelity simulation manikin higher than those who perform the practice with the standard demonstration method?
* Are the satisfaction levels of nursing students who perform the simulation practice with the scenario-based high-fidelity simulation manikin higher than those who perform the practice with the standard demonstration method? Researchers will compare two groups of nursing students training with high-fidelity simulation manikin and training with standard demonstration method.

ELIGIBILITY:
Inclusion Criteria:

* First-year nursing students
* Not have been trained in simulation before
* Taking a nursing fundamentals course for the first time
* Open to communication and volunteering to be involved in the study

Exclusion Criteria:

* Not meeting the inclusion criteria
* Not volunteering to participate in the study

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Assessing nursing students of skills in wearing-removing personal protective equipment | 1 month
  Procedural Steps Checklist was used to assess nursing wearing-removing skills. The checklist for PPE wearing-removal skills was created by the researchers based on their review of the relevant literature (Göçmen Baykara et al. 2020; Patricia Potter et al. 2020; World Health Organization 2021). Opinions were received from five faculty members with expertise in Fundamentals of Nursing for the checklist, and Kendall's W coefficient for the checklist was found as 0.776 (p < .001). The Cronbach's alpha coefficient of the checklist was calculated as 0.64, which showed a moderate level of internal consistency. The checklist to be used for assessment was finalized, and it consisted of 17 items. Each item was scored as 0 or 1, and the minimum and maximum total scores of the checklist were 0 and 17. When the participant performed the procedural step, they received 1 point for the related item, while they received 0 points when they failed to perform the step.
Describing nursing students of satisfaction levels | 1 month
  VAS was used to determine which model was more satisfactory to nursing students. VAS was used to measure the satisfaction levels of the participants based on their own assessment between "0 (not satisfied at all) and 10 (very satisfied)".

SECONDARY OUTCOMES:
Establish fear of COVID-19 levels of nursing students | Through study completion, an average of 1 month
  Fear of COVID-19 Scale (FCV-19S) was used to determine the COVID-19 fear levels of nursing students. This scale, which was developed by Ahorsu et al. (2020), was adapted to Turkish culture by Bakioğlu, Korkmaz, and Ercan (2020). It is a unidimensional scale consisting of seven items. The item-total correlation coefficients of the scale were reported to vary from 0.47 to 0.56, while its factor loads were reported to vary from 0.66 to 0.74. The Cronbach's alpha coefficient of the scale was reported as α = 0.82. A set of validity and reliability analyses was carried out for the five-point Likert-type scale in its Turkish adaptation study. The authors conducting the study reported Cronbach's alpha coefficient of the scale as 0.88. Other authors also adapted the scale to Turkish (Satıcı et al. 2020). Considering the results of adaptation studies, it may be stated that it is a valid and reliable scale (Ahorsu et al. 2022; Bakioğlu, Korkmaz, and Ercan 2021).

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Planning to make a manuscript for this study and sharing participant identification information and outcomes.

REFERENCES:
- [Background] Koukourikos K, Tsaloglidou A, Kourkouta L, Papathanasiou IV, Iliadis C, Fratzana A, Panagiotou A. Simulation in Clinical Nursing Education. Acta Inform Med. 2021 Mar;29(1):15-20. doi: 10.5455/aim.2021.29.15-20. PMID 34012208
- [Background] Ahorsu DK, Lin CY, Imani V, Saffari M, Griffiths MD, Pakpour AH. The Fear of COVID-19 Scale: Development and Initial Validation. Int J Ment Health Addict. 2022;20(3):1537-1545. doi: 10.1007/s11469-020-00270-8. Epub 2020 Mar 27. PMID 32226353
- [Background] Kuru Alici N, Ozturk Copur E. Anxiety and fear of COVID-19 among nursing students during the COVID-19 pandemic: A descriptive correlation study. Perspect Psychiatr Care. 2022 Jan;58(1):141-148. doi: 10.1111/ppc.12851. Epub 2021 May 20. PMID 34018195
- [Background] Alsolais A, Alquwez N, Alotaibi KA, Alqarni AS, Almalki M, Alsolami F, Almazan J, Cruz JP. Risk perceptions, fear, depression, anxiety, stress and coping among Saudi nursing students during the COVID-19 pandemic. J Ment Health. 2021 Apr;30(2):194-201. doi: 10.1080/09638237.2021.1922636. Epub 2021 May 12. PMID 33978543
- [Background] Apisarnthanarak A, Apisarnthanarak P, Siripraparat C, Saengaram P, Leeprechanon N, Weber DJ. Impact of anxiety and fear for COVID-19 toward infection control practices among Thai healthcare workers. Infect Control Hosp Epidemiol. 2020 Sep;41(9):1093-1094. doi: 10.1017/ice.2020.280. Epub 2020 Jun 8. No abstract available. PMID 32507115
- [Background] Bakioglu F, Korkmaz O, Ercan H. Fear of COVID-19 and Positivity: Mediating Role of Intolerance of Uncertainty, Depression, Anxiety, and Stress. Int J Ment Health Addict. 2021;19(6):2369-2382. doi: 10.1007/s11469-020-00331-y. Epub 2020 May 28. PMID 32837421
- [Background] Basak T, Unver V, Moss J, Watts P, Gaioso V. Beginning and advanced students' perceptions of the use of low- and high-fidelity mannequins in nursing simulation. Nurse Educ Today. 2016 Jan;36:37-43. doi: 10.1016/j.nedt.2015.07.020. Epub 2015 Jul 29. PMID 26282193
- [Background] Bouchoucha SL, Phillips NM, Lucas J, Kilpatrick M, Hutchinson A. An investigation into nursing students' application of infection prevention and control precautions. Nurse Educ Today. 2021 Sep;104:104987. doi: 10.1016/j.nedt.2021.104987. Epub 2021 May 29. PMID 34098422
- [Background] Campanati FLDS, Ribeiro LM, Silva ICRD, Hermann PRS, Brasil GDC, Carneiro KKG, Funghetto SS. Clinical simulation as a Nursing Fundamentals teaching method: a quasi-experimental study. Rev Bras Enferm. 2021 Oct 18;75(2):e20201155. doi: 10.1590/0034-7167-2020-1155. eCollection 2021. English, Portuguese. PMID 34669900
- [Background] Cheng A, Kessler D, Mackinnon R, Chang TP, Nadkarni VM, Hunt EA, Duval-Arnould J, Lin Y, Cook DA, Pusic M, Hui J, Moher D, Egger M, Auerbach M; International Network for Simulation-based Pediatric Innovation, Research, and Education (INSPIRE) Reporting Guidelines Investigators. Reporting guidelines for health care simulation research: extensions to the CONSORT and STROBE statements. Adv Simul (Lond). 2016 Jul 25;1:25. doi: 10.1186/s41077-016-0025-y. eCollection 2016. PMID 29449994
- [Background] Driscoll B, Evans D. Nursing Infection Control Practice Adherence, Related Barriers, and Methods of Intervention. J Nurs Adm. 2022 Mar 1;52(3):132-137. doi: 10.1097/NNA.0000000000001120. PMID 35170577
- [Background] Elo S, Kyngas H. The qualitative content analysis process. J Adv Nurs. 2008 Apr;62(1):107-15. doi: 10.1111/j.1365-2648.2007.04569.x. PMID 18352969
- [Background] Eyikara E, Baykara ZG. Effect of simulation on the ability of first year nursing students to learn vital signs. Nurse Educ Today. 2018 Jan;60:101-106. doi: 10.1016/j.nedt.2017.09.023. Epub 2017 Oct 13. PMID 29078202
- [Background] Fawaz MA, Hamdan-Mansour AM. Impact of high-fidelity simulation on the development of clinical judgment and motivation among Lebanese nursing students. Nurse Educ Today. 2016 Nov;46:36-42. doi: 10.1016/j.nedt.2016.08.026. Epub 2016 Aug 25. PMID 27591378
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Lei YY, Zhu L, Sa YTR, Cui XS. Effects of high-fidelity simulation teaching on nursing students' knowledge, professional skills and clinical ability: A meta-analysis and systematic review. Nurse Educ Pract. 2022 Mar;60:103306. doi: 10.1016/j.nepr.2022.103306. Epub 2022 Feb 2. PMID 35202957
- [Background] Medina Fernandez IA, Carreno Moreno S, Chaparro Diaz L, Gallegos-Torres RM, Medina Fernandez JA, Hernandez Martinez EK. Fear, Stress, and Knowledge regarding COVID-19 in Nursing Students and Recent Graduates in Mexico. Invest Educ Enferm. 2021 Feb;39(1):e05. doi: 10.17533/udea.iee.v39n1e05. PMID 33687809
- [Background] Najjar RH, Lyman B, Miehl N. Nursing students' experiences with high-fidelity simulation. Int J Nurs Educ Scholarsh. 2015 Mar 19;12:/j/ijnes.2015.12.issue-1/ijnes-2015-0010/ijnes-2015-0010.xml. doi: 10.1515/ijnes-2015-0010. PMID 25803087
- [Background] Padilha JM, Machado PP, Ribeiro A, Ramos J, Costa P. Clinical Virtual Simulation in Nursing Education: Randomized Controlled Trial. J Med Internet Res. 2019 Mar 18;21(3):e11529. doi: 10.2196/11529. PMID 30882355
- [Background] Pol-Castaneda S, Carrero-Planells A, Moreno-Mulet C. Use of simulation to improve nursing students' medication administration competence: a mixed-method study. BMC Nurs. 2022 May 16;21(1):117. doi: 10.1186/s12912-022-00897-z. PMID 35578199
- [Background] Tabah A, Ramanan M, Laupland KB, Buetti N, Cortegiani A, Mellinghoff J, Conway Morris A, Camporota L, Zappella N, Elhadi M, Povoa P, Amrein K, Vidal G, Derde L, Bassetti M, Francois G, Ssi Yan Kai N, De Waele JJ; PPE-SAFE contributors. Personal protective equipment and intensive care unit healthcare worker safety in the COVID-19 era (PPE-SAFE): An international survey. J Crit Care. 2020 Oct;59:70-75. doi: 10.1016/j.jcrc.2020.06.005. Epub 2020 Jun 13. PMID 32570052
- [Background] Verbeek JH, Rajamaki B, Ijaz S, Sauni R, Toomey E, Blackwood B, Tikka C, Ruotsalainen JH, Kilinc Balci FS. Personal protective equipment for preventing highly infectious diseases due to exposure to contaminated body fluids in healthcare staff. Cochrane Database Syst Rev. 2020 Apr 15;4(4):CD011621. doi: 10.1002/14651858.CD011621.pub4. PMID 32293717
- [Background] Watson C, Gomez-Ibanez R, Granel N, Bernabeu-Tamayo MD. Nursing students first experience on high fidelity simulation: A phenomenological research study. Nurse Educ Pract. 2021 Aug;55:103162. doi: 10.1016/j.nepr.2021.103162. Epub 2021 Jul 23. PMID 34332280
- [Background] Yu M, Yang MR. Effectiveness and Utility of Virtual Reality Infection Control Simulation for Children With COVID-19: Quasi-Experimental Study. JMIR Serious Games. 2022 May 27;10(2):e36707. doi: 10.2196/36707. PMID 35575818
- See also: Reference — https://dergipark.org.tr/tr/download/issue-full-file/69367
- See also: Reference — https://doi.org/10.1016/j.ecns.2018.05.001
- See also: Reference — https://www.inacsl.org/healthcare-simulation-standards